CLINICAL TRIAL: NCT01221805
Title: STA®-Liatest®D-Di-Exclusion of Venous Thromboembolism
Acronym: DiET
Status: Completed | Type: Observational
Sponsor: Diagnostica Stago (Industry)
Collaborators: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Other Study IDs: DCIC 10 18
Record Dates: First submitted 2010-10-12; First posted 2010-10-15 (Estimated); Last update posted 2016-08-05 (Estimated); Status verified 2016-08

CONDITIONS: Deep Venous Thrombosis; Pulmonary Embolism; D-dimer
Keywords: deep venous thrombosis; pulmonary embolism; venous thromboembolism; D-dimer; Wells score; Wells clinical pretest probability
MeSH Terms: conditions — Venous Thrombosis; Pulmonary Embolism; Venous Thromboembolism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — plasma samples (at least 1 aliquot 0.5 ml) will be collected at the initial visit of patients with low or moderate PTP
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to demonstrate the ability of STA® Liatest® D-Di combined with a clinical pretest probability (PTP) to safely exclude pulmonary embolism (PE) or Deep Venous Thrombosis (DVT) in a 3 month follow-up.

DETAILED DESCRIPTION:
The study population will be selected from prospective, consecutive ambulatory outpatients suspected of having venous thromboembolism.

These patients will first be evaluated using the Wells score:

* patients with low or moderate pretest probability will be considered for D-dimer testing, those with D-dimer positive will be considered for an imaging procedure,
* patients with high pretest probability will be considered for an imaging procedure.

Patients with "low or moderate" pretest probability and a negative D-Dimer result will be followed for 3 months to evaluate potential development of deep venous thrombosis and/or pulmonary embolism.

These patients will be contacted by phone 3 month after their first visit.

ELIGIBILITY:
INCLUSION CRITERIA

1. Patient is < 80 years old.
2. Patient presenting at least one of these symptoms indicative of proximal DVT or PE:

   * symptoms for proximal DVT: leg pain, tenderness (discomfort through palpation), leg swelling, and /or edema,
   * symptoms for PE: hemoptysis, lung related chest pain, dyspnea.
3. Patient provides written informed consent to participate in the study (or verbal no-opposition, as allowed by local regulations)
4. Patient is willing to comply with specified follow-up evaluation at 3 months and can be contacted by telephone

EXCLUSION CRITERIA

1. Patient presenting with a condition that may be associated with increased D-dimer levels, even in the absence of VTE, such as:

   * Fibrinolytic therapy within the previous seven (7) days,
   * Bone fracture or surgery (with general anesthesia longer than thirty (30) minutes) within the previous one (1) month,
   * Deep hematoma diagnosed by imaging techniques within the previous one (1) month,
   * Disseminated malignancies and active cancer (active cancer defined as: cancer for which therapeutic or palliative treatment is either ongoing at the time of enrolment or has stopped less than six (6) months before enrolment),
   * Sepsis, severe infections, pneumonia within the previous 1 month,
   * Known liver cirrhosis,
   * Pregnancy or post-partum within the previous 1 month,
   * Atherosclerotic vascular disease thrombosis within the previous 1month (e.g. myocardial infarction, stroke, coronary syndrome, peripheral artery disease stage III or IV),
   * Sickle cell disease,
2. Patients presenting with a suspect thrombotic event related to catheter implantation
3. Ongoing therapeutic anticoagulants (curative and preventive treatment) starting twenty four (24) hours or more before the D-dimer is measured
4. Previous anticoagulant therapy stopped less than three (3) months before the D-dimer is measured
5. Patients with previous DVT/PE occurred less than three (3) months from screening.
6. Suspect thrombotic events in other locations at screening, including distal to the knee and upper extremity DVT (based on standard of care examinations)
7. Patients with known tissue plasminogen activator (tPA) deficiency
8. Patient participating or who has participated within one month of enrollment in another investigational study
9. Major co-morbid condition(s) or other reasons that could limit the patient's ability to participate in the study or to comply with follow-up requirements, or impact the scientific integrity of the study

Max Age: 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population will be recruited from prospective, consecutive, ambulatory outpatients (presenting at the emergency unit or outpatient clinic) suspected of having venous thromboembolism
Sampling Method: Non-Probability Sample
Enrollment: 2040 (Actual)
Dates: Start 2011-11; Primary Completion 2016-03 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
To demonstrate the ability of STA Liatest DDi combined with a clinical pretest probability (PTP) to safely exclude pulmonary embolism or deep venous thrombosis in a 3 month follow-up | at 3 months
  Occurence of pulmonary embolism or deep venous thrombosis during the 3 month follow-up after negative diagnosis (i.e. patients with PTP low/moderate and negative STA Liatest D-Di test)

SECONDARY OUTCOMES:
1. To analyse results homogeneity (inter-centers) in the group "positive D-dimer result and negative diagnosis" (descriptive statistics only). 2. To determine prevalence of VTE in PTP high patients based on imaging results | at 3 months
  1. Prevalence of VTE in PTP high patients based on imaging results.

CONTACTS AND LOCATIONS:
Overall Officials: GILLES PERNOD, MD PhD, Principal Investigator — University Hospital, Grenoble
Locations (18):
- United States (11):
  - Northwestern Medical Center, Chicago, Illinois
  - Indiana University Health, Indianapolis, Indiana
  - University of Iowa, Iowa City, Iowa
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham and Woman's Hosp, Boston, Massachusetts
  - Moses Cone Memorial Hospital, Greensboro, North Carolina
  - Univeristy Medical Center, Colombus, Ohio
  - Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Lehigh Valley Hospital Health Network, Allentown, Pennsylvania
  - Medical Center of South Carolina, Charleston, South Carolina
  - Texas Health Fort Worth Hospital, Fort Worth, Texas
- Maisonneuve Rosemont Hospital, Montreal, Canada
- France (2):
  - University Hospital, Dijon
  - University Hospital, Grenoble
- Italy (2):
  - University Hospital, Bologna
  - IRCCS H San Raffaele, Milan
- Spain (2):
  - University Hospital, Alicante
  - General Hospital, Soria

REFERENCES:
- [Background] Keeling DM, Mackie IJ, Moody A, Watson HG; Haemostasis and Thrombosis Task Force of the British Committee for Standards in Haematology. The diagnosis of deep vein thrombosis in symptomatic outpatients and the potential for clinical assessment and D-dimer assays to reduce the need for diagnostic imaging. Br J Haematol. 2004 Jan;124(1):15-25. doi: 10.1046/j.1365-2141.2003.04723.x. No abstract available. PMID 14675404
- [Background] Goekoop RJ, Steeghs N, Niessen RW, Jonkers GJ, Dik H, Castel A, Werker-van Gelder L, Vlasveld LT, van Klink RC, Planken EV, Huisman MV. Simple and safe exclusion of pulmonary embolism in outpatients using quantitative D-dimer and Wells' simplified decision rule. Thromb Haemost. 2007 Jan;97(1):146-50. PMID 17200782
- [Background] Kelly J, Hunt BJ. A clinical probability assessment and D-dimer measurement should be the initial step in the investigation of suspected venous thromboembolism. Chest. 2003 Sep;124(3):1116-9. No abstract available. PMID 12970044
- [Background] Pasha SM, Klok FA, Snoep JD, Mos IC, Goekoop RJ, Rodger MA, Huisman MV. Safety of excluding acute pulmonary embolism based on an unlikely clinical probability by the Wells rule and normal D-dimer concentration: a meta-analysis. Thromb Res. 2010 Apr;125(4):e123-7. doi: 10.1016/j.thromres.2009.11.009. Epub 2009 Nov 26. PMID 19942258
- [Background] Perrier A, Desmarais S, Goehring C, de Moerloose P, Morabia A, Unger PF, Slosman D, Junod A, Bounameaux H. D-dimer testing for suspected pulmonary embolism in outpatients. Am J Respir Crit Care Med. 1997 Aug;156(2 Pt 1):492-6. doi: 10.1164/ajrccm.156.2.9702032. PMID 9279229
- [Background] Wells PS, Anderson DR, Rodger M, Forgie M, Kearon C, Dreyer J, Kovacs G, Mitchell M, Lewandowski B, Kovacs MJ. Evaluation of D-dimer in the diagnosis of suspected deep-vein thrombosis. N Engl J Med. 2003 Sep 25;349(13):1227-35. doi: 10.1056/NEJMoa023153. PMID 14507948
- [Derived] Pernod G, Caterino J, Maignan M, Tissier C, Kassis J, Lazarchick J; DIET study group. D-Dimer Use and Pulmonary Embolism Diagnosis in Emergency Units: Why Is There Such a Difference in Pulmonary Embolism Prevalence between the United States of America and Countries Outside USA? PLoS One. 2017 Jan 13;12(1):e0169268. doi: 10.1371/journal.pone.0169268. eCollection 2017. PMID 28085911